CLINICAL TRIAL: NCT02190929
Title: Educational Needs of Patients With Systemic Vasculitis- an International Survey
Brief Title: Educational Needs of Patients With Systemic Vasculitis
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Boston University (Other); University of Pennsylvania (Other); Data Management and Coordinating Center (DMCC) (Other)
Responsible Party: Sponsor
Other Study IDs: 5534
Record Dates: First submitted 2014-05-30; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Behcet's Disease; Churg-Strauss Syndrome; Vasculitis, Central Nervous System; Giant Cell Arteritis; Wegener Granulomatosis; Henoch-Schoenlein Purpura; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu's Arteritis
MeSH Terms: conditions — Behcet Syndrome; Churg-Strauss Syndrome; Vasculitis, Central Nervous System; Giant Cell Arteritis; Granulomatosis with Polyangiitis; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vasculitis Contact Registry Patients: Patients will be recruited from within the Vasculitis Clinical Research Consortium (VCRC) Patient Contact Registry to participate in an online questionnaire. More than 3000 patients, representing all the different types of idiopathic vasculitis, are currently enrolled into the on-line registry. The different types of vasculitis available for study include: Behçets disease, Churg-Strauss Syndrome, CNS Vasculitis, Giant Cell Arteritis, granulomatosis with polyangiitis (Wegener's granulomatosis), Henoch-Schöenlein Purpura, Microscopic Polyangiitis, Polyarteritis Nodosa, or Takayasu's Arteritis.

SUMMARY:
A cross-sectional study design and online questionnaire was used to assess the informational needs of patients with several different types of systemic vasculitis. Patients were recruited from within the Vasculitis Clinical Research Consortium (VCRC) online Patient Contact Registry1. Survey responses from participants in the VCRC Patient Contact Registry were compared to responses from a similar survey recently administered to patients within a United Kingdom (UK) based vasculitis support group (Vasculitis UK).

DETAILED DESCRIPTION:
All patients enrolled in the Vasculitis Clinical Research Consortium's Contact Registry were invited via email to participate in this study. The Contract Registry includes people who self-identify as having one of the following types of vasculitis: Behçets disease, Churg-Strauss Syndrome, CNS Vasculitis, Giant Cell Arteritis, granulomatosis with polyangiitis (Wegener's granulomatosis), Henoch-Schöenlein Purpura, Microscopic Polyangiitis, Polyarteritis Nodosa, or Takayasu's Arteritis. People voluntarily enroll in this Registry with the understanding that they will receive information about clinical studies for which they might be eligible. The introductory email included basic information about the study and all of the required elements for informed consent in a brief format. Once participants agreed to participate in the study, they were directed to the online questionnaire.

When completing the questionnaire, the patients were asked a series of questions. The questionnaire content was included as an appendix. The online questionnaire version was thoroughly tested for usability.

It was expected that most participants wouldrequire approximately 10-15 minutes to complete the questionnaire.

The survey data is stored by the Rare Diseases Clinical Research Network Data Management and Coordinating Center (DMCC) at the University of South Florida. The data is de-identified. Names or other personal health information were not collected.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the VCRC Contact Registry
* Patient reported diagnosis of Behçets disease, Churg-Strauss Syndrome, CNS Vasculitis, Giant Cell Arteritis, granulomatosis with polyangiitis (Wegener's granulomatosis), Henoch-Schöenlein Purpura, Microscopic Polyangiitis, Polyarteritis Nodosa, Takayasu's Arteritis.
* 18 years of age or older
* English speaking

Exclusion Criteria:

* Inability to provide informed consent and complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from within the Vasculitis Clinical Research Consortium (VCRC) Patient Contact Registry to participate in an online questionnaire. More than 3000 patients, representing all the different types of idiopathic vasculitis, are currently enrolled into the on-line registry. The different types of vasculitis available for study include: Behçets disease, Churg-Strauss Syndrome, CNS Vasculitis, Giant Cell Arteritis, granulomatosis with polyangiitis (Wegener's granulomatosis), Henoch-Schöenlein Purpura, Microscopic Polyangiitis, Polyarteritis Nodosa, or Takayasu's Arteritis.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Preferred method and component of education materials for patients with vasculitis | Up to 24 months from the last patient assessment received
  The outcome measure will be evaluated based on the cross-sectional online questionnaire. The questionnaire is the only study procedure for this online patient contact registry protocol and will be the sole analysis tool for the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Watts, DM, Study Chair — University of East Anglia; Janice Mooney, M.Sc., Study Chair — University of East Anglia; Peter C. Grayson, MD, Study Chair — Boston University; Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania; Amanda M. Terry, MA, Study Chair — University of South Florida College of Medicine
Locations (1):
- University of South Florida Data Management Coordinating Center, Tampa, Florida, United States